CLINICAL TRIAL: NCT06842407
Title: Nuovi Bersagli Per lo Sviluppo di Anticorpi Monoclonali Per Immunoterapia - (Novel Targets for the Development of Monoclonal Antibodies for Immunotherapy)
Brief Title: Novel Targets for the Development of Monoclonal Antibodies for Immunotherapy)
Acronym: Immuno-ab
Status: Recruiting | Type: Observational
Sponsor: Checkmab S.r.l. (Industry)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: ID3411
Record Dates: First submitted 2025-02-14; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Healthy Donors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma Frozen cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Donors: subjects over 18 years of age

SUMMARY:
The first objective of the project consists in the preclinical validation of new possible molecular targets associated with intratumoral T regulatory cells. The second objective consists in the selection of monoclonal antibodies with therapeutic potential, specific for the selected targets.

ELIGIBILITY:
Inclusion Criteria:

* blood donors
* age of 18 years or more
* able to sign informed consent

Exclusion Criteria:

* age below 18 years
* Positive for HIV, HCV, HBV
* not suitable for blood donation
* not able to understand or sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Validation of molecular targets for immunotherapy | 04.2023-06.2026
Selection of therapeutic antibodies | 04.2023-06.2026

SECONDARY OUTCOMES:
Set up of immunological assays to adress monoclonal antibodies mechanism of action | 04.2023-06.2026

CONTACTS AND LOCATIONS:
Locations (1):
- S.C. Medicina Trasfusionale - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy